CLINICAL TRIAL: NCT00288288
Title: Prospective Registry of Epicardial LV Leads Placed During Cardiac Surgery Procedures
Status: Completed | Type: Observational
Sponsor: University of Kansas (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Loren Berenbom, MD, Principal Investigator, University of Kansas
Organization: University of Kansas Medical Center (Other)
Other Study IDs: PROPEL
Record Dates: First submitted 2006-02-03; First posted 2006-02-07 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Epicardial left ventricular lead placement during a clinically indicated open chest surgery
  Interventions: Procedure: Epicardial left ventricular lead placement
- 2: Transvenous left ventricular lead implant during a clinically indicated CRT system implant
  Interventions: Procedure: Transvenous left ventricular lead implant

INTERVENTIONS:
Procedure: Epicardial left ventricular lead placement — Epicardial left ventricular lead placement
  Groups: 1
Procedure: Transvenous left ventricular lead implant — Transvenous left ventricular lead implant
  Groups: 2

SUMMARY:
The primary purpose of this study is to compare the time, risk and cost savings of 2 patient groups who receive FDA approved left ventricular pacing leads.

DETAILED DESCRIPTION:
The purpose of this study is to: a) examine the usefulness of placing an epicardial LV lead at the time of open chest surgery in patients who are likely to benefit from a CRT system following their surgery; b) compare differences between patients who receive LV leads using the transvenous approach and those patients who receive LV leads using the epicardial approach; and c) assess the cost effectiveness of placing the LV lead via the transvenous versus the epicardial approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Left ventricular ejection fraction < or = 35%
2. QRS duration greater than or = to 120ms
3. NYHA Functional Class 3 or 4
4. Age > or = to 18 years

Exclusion Criteria:

1. No previous pacemaker or ICD implant
2. No permanent atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2006-03; Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loren Berenbom, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States